CLINICAL TRIAL: NCT03535116
Title: The Effect of Intra-operative Ketorolac on Hematoma Rates in Breast Reduction Surgery: A Double Blind Randomized Control Trial
Brief Title: The Effect of Intra-operative Ketorolac on Hematoma Rates in Breast Reduction Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Chandran Medical Prof Corp (Other)
Responsible Party: Principal Investigator, Geethan Chandran, Assistant Professor, Dr. Chandran Medical Prof Corp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 33
Record Dates: First submitted 2018-05-13; First posted 2018-05-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hematoma Postoperative
MeSH Terms: interventions — Ketorolac; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double Blind Randomized Control Trial of breast reduction patients and their postoperative hematoma rates with the use of ketorolac
Who Masked: Participant, Care Provider
Masking Description: drug vs placebo(saline). Identification is in a sealed envelope. The anesthetist gives the medication without telling the surgeon or the patient what medication is given(patient will be under a general anesthetic). Neither patient or surgeon will know what the patient gets until the follow up period(6 weeks) is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving ketorolac (Experimental): Patient receives 30mg IV ketorolac(single dose) towards the end of the operation.
  Interventions: Drug: Ketorolac
- Control (Placebo Comparator): Patients receive saline intravenously towards the end of the operation.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketorolac — Toradol is a type of brand name. We will be using the generic version.
  Arms: Patients receiving ketorolac
Drug: Saline — injectable normal saline
  Arms: Control

SUMMARY:
It has been a longstanding teaching in plastic surgery that intra-operative ketorolac use for postoperative pain control increases hematoma and bleeding in breast reduction surgery. However, there is no literature that supports this teaching. Ketorolac is used routinely in free flap reconstruction including breast reconstruction as well as many other surgeries including hand surgery without increased risks of hematoma or bleeding. Ketorolac has been shown to give good postoperative pain control. The object of this study is to look at whether ketorolac increases the rate of hematoma/bleeding in breast reduction. If there is no increased risk of hematoma, then ketorolac can be used safely for postoperative pain control with an increased risk of hematoma/bleeding. Normally, without using ketorolac, the hematoma rates in a breast reduction are 1-2%.

DETAILED DESCRIPTION:
STUDY PROTOCOL

The Effect of Intra-operative Ketorolac on Hematoma Rates in Breast Reduction Surgery: A Double Blind Randomized Control Trial

Purpose: The purpose of this study to investigate hematoma rates of a single dose of ketorolac given intra-operatively in breast reduction surgery.

Hypothesis: There is no statistically significant difference between the ketorolac and placebo in hematoma rates after intra-operative single use in breast reduction surgery.

PROTOCOL

A Power analysis and sample size estimation was carried out with an alpha=0.05 and a beta=0.80. This gave the study a power of 0.94 and sample size estimation of 260 patients per group.

A consent form will be developed and the University of Saskatchewan ethics approval will be obtained. The study will be registered as a trial through ClinicalTrials.gov.

The plastic surgeons in the study will start recruiting patients during their initial consultation for breast reduction. The consultation will determine if the patient is a candidate for a breast reduction clinically. The candidacy for a breast reduction is determined strictly on a clinical basis and only then the patient will be considered to participate in the study. If the patient meets inclusion criteria, the patient will be asked to participate in the study. The process of the study as it pertains to the patient and the risks/benefits of the study and the study medication will be discussed with the patient by the surgeon.

If the patient agrees to participate in the study, they will be asked to sign the consent form on the day of surgery. They will have a patient number(1-260) assigned to them. A computer generated randomization process will determine if the patient will get ketorolac or saline(placebo). A small piece of paper with either of the words "ketorolac" or "saline" will be placed in an envelope with the corresponding patient number and sealed. This randomization and envelope will be administered by the clinic nurse and a computer spreadsheet of the patient number and medication to administered will be kept by the clinic nurse. The surgeon or patient will not have knowledge of this.

The breast reduction surgery will be performed in the usual manner as clinically dictated. The anesthetist will be given the sealed envelope at the beginning of the case. Towards the end of the operation, the anesthetist will open the envelope and administer the medication as indicated in the content of the envelope, reseal the envelope and record what was given on their anesthetic record. The surgeon will not have any knowledge of what medication was administered.

After the breast reduction is finished, the patient will be transferred to the recovery room. The surgeon will examine the patient in the recovery room or day surgery before the patient is discharged to determine if there is a hematoma. If there is a hematoma, the surgeon will inform the clinic nurse of such and the treatment of the hematoma(eg. Re-operation, observation etc). Before the patient is discharged, the day surgery nurse will ask the patient to indicate on the visual analog scale about their pain level(scale of 1-10). Then the patient will be discharged home if appropriate. The patient will have instructions on the signs of hematoma to watch out for in the form of written instructions.

Two weeks postoperatively and 6 weeks postoperatively, the patient will be seen for a followup by the clinic nurse as an independent assessor for a hematoma. The presence or absence of a hematoma will be recorded. If there is a hematoma, the surgeon will be notified to assess the patient. The treatment of the hematoma will be communicated to the clinic nurse by the surgeon.

After the 6 week followup, the study for that patient will be finished. If the patient wishes to know what medication that they received intra-operatively, the clinic nurse can inform them at that point.

All data will be stored in a password protected computer at Dr. Chandran's office at 210-206 Wellman Crescent, Saskatoon, Saskatchewan, Canada. At no point will any of the identifiable data in this study's database be transferred off the premises.

After the collection of data for all patients, the data will be analyzed by the statistician for the Department of Surgery of the University of Saskatchewan or their equivalent. The data will be de-identified of patient names before sending to the statistician. A master list with the patient names and the corresponding patient number will only be kept at Dr. Chandran's office(above). The results will be discussed by the research team and publication/presentation shall be determined.

ELIGIBILITY:
Inclusion Criteria:

Age > 18

* female
* clinically met criteria for breast reduction(large heavy breasts)

Exclusion Criteria:

* smokers
* morbid obesity
* history of kidney failure
* allergy to non steroidal anti-inflammatories
* did not wish or unable to consent to be in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — must be female as these are surgeries for breast reductions
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematoma | 6 weeks
  Postoperative hematoma

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No